CLINICAL TRIAL: NCT06488339
Title: Efficacy and Safety of Food Replacement on Weight Control in Overweight Volunteers
Brief Title: Food Replacement on Weight Control in Overweight Volunteers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Collaborators: Mae Fah Luang University (Other)
Responsible Party: Principal Investigator, Pornanong Aramwit, Pharm.D., Ph.D, Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: EC23238-20
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Weight Gain
MeSH Terms: conditions — Weight Gain | interventions — Proteins

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protein and oil supplement (Experimental): Take 1 sachet/day replaced dinner
  Interventions: Dietary Supplement: Protein and oil supplement
- Normal dietary meal (No Intervention): Take normal dietary meal for dinner

INTERVENTIONS:
Dietary Supplement: Protein and oil supplement — Take 1 sachet/day replaced dinner
  Arms: Protein and oil supplement

SUMMARY:
Volunteers will be divided into two groups which are protein and oil supplement group and normal dietary group. For protein and oil supplement group, they will take 1 sachet of product replaced dinner every day for 8 weeks. For normal dietary group, they will take regular dinner every day for 8 weeks. Weight, body mass index, body composition, waist and hip circumference, skin fold thickness, and chemistry in blood will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* Body mass index more than 23 kg/m2
* No heart disease, diabetes mellitus, thyroid disease, cancer, liver and kidney diseases
* Wiling to attend the study

Exclusion Criteria:

* Allergic to protein, grains, guar gum
* Take medicine, supplement, herbal substance for weight control within 1 month
* During intermittent fasting
* Take birth control pill, steroids, anti-depressant drugs, and anti-epilepsy drugs
* Cushing syndrome's
* Pregnancy and lactation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Weight | 8 weeks
  Weight of volunteers (kg)

SECONDARY OUTCOMES:
Body mass index | 8 weeks
  Body mass index of volunteers (kg/m2)
Percentage of body fat | 8 weeks
  Percentage of body fat (%) using bioelectrical impedance analysis (BIA)
Percentage of visceral fat | 8 weeks
  Percentage of visceral fat (%) using bioelectrical impedance analysis (BIA)
Percentage of subcutaneous fat | 8 weeks
  Percentage of subcutaneous fat (%) using bioelectrical impedance analysis (BIA)
Percentage of muscle | 8 weeks
  Percentage of muscle (%) using bioelectrical impedance analysis (BIA)
Waist Circumference | 8 weeks
  Waist Circumference (cm)
Hip Circumference | 8 weeks
  Hip Circumference (cm)
Skin fold thickness | 8 weeks
  Skin fold thickness (mm) using Skinfold Caliper
Total cholesterol | 8 weeks
  Blood total cholesterol (mg/dL)
Low density lipoprotein | 8 weeks
  Low density lipoprotein (mg/dL) in blood
High density lipoprotein | 8 weeks
  High density lipoprotein (mg/dL) in blood
Triglycerides | 8 weeks
  Triglycerides (mg/dL) in blood
Fasting blood sugar | 8 weeks
  Fasting blood sugar (mg/dL) in blood
Hemoglobin A1C | 8 weeks
  Hemoglobin A1C (%) in blood
Total protein | 8 weeks
  Total protein (g/dL) in blood
Hemoglobin | 8 weeks
  Hemoglobin (g/dL) in blood
SIRT1 (NAD-dependent deacetylase sirtuin-1) | 8 weeks
  SIRT1 (NAD-dependent deacetylase sirtuin-1) (%) in blood
8-hydroxy-2-deoxyguanosine | 8 weeks
  8-hydroxy-2-deoxyguanosine (%) in blood
Blood urea nitrogen | 8 weeks
  Blood urea nitrogen (mg/dL) in blood
Creatinine | 8 weeks
  Creatinine (mg/dL) in blood
Aspartate transaminase | 8 weeks
  Aspartate transaminase (U/L) in blood
Alanine aminotransferase | 8 weeks
  Alanine aminotransferase (U/L) in blood
Alkaline phosphatase | 8 weeks
  Alkaline phosphatase (U/L) in blood